CLINICAL TRIAL: NCT06113861
Title: Diagnostic Innovations for Pediatric Tuberculosis in Bolivia
Status: Recruiting | Type: Observational
Sponsor: Tulane University (Other)
Collaborators: Asociacion Benefica Prisma (Other); Universidad Peruana Cayetano Heredia (Other); Johns Hopkins Bloomberg School of Public Health (Other)
Responsible Party: Principal Investigator, Richard A. Oberhelman, Professor, Tulane University
Other Study IDs: R01AI173021 (NIH)
Record Dates: First submitted 2023-10-27; First posted 2023-11-02 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-09

CONDITIONS: Tuberculosis
Keywords: Diagnostic testing; Children; Imaging analysis
MeSH Terms: conditions — Tuberculosis | interventions — AIDS Serodiagnosis; Diagnostic Imaging

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Months
Biospecimen Retention: Samples With DNA — Plasma samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Presumptive pediatric TB cases-- Test population: Inclusion criteria: Children ages 2 months to 14 years with symptomatic disease and suspicion of TB (based on Bolivian Ministry of Health guidelines).
  Exclusion criteria (prior treatment for TB in 12 mo, current treatment for TB, weight < 2.5 kg., instability, positive COVID-19 test) Study subgroups are determined in part based on the results of diagnostic tests and on clinical response.
  A. Confirmed TB
  * Symptomatic by case definition from the 2015 NIH Expert Panel
  * Positive culture or positive Xpert MTB/RIF from at least one sample.
  B. Unconfirmed TB-
  * Symptomatic and clinical/radiographic evaluation consistent with TB, by case definition from the 2015 NIH Expert Panel
  * Negative M. tuberculosis culture and negative Xpert MTB/RIF from all samples.
  C. Unlikely TB---
  * Symptomatic BUT clinical/radiographic eval does NOT meet criteria for Unconfirmed TB, per clinical definition-2015 Expert Panel
  * Negative culture and negative Xpert MTB/RIF from all specimens.
  Interventions: Diagnostic Test: Quantiferon Gold; Diagnostic Test: HIV serology; Diagnostic Test: Respiratory secretion culture (sputum or gastric aspirate_; Diagnostic Test: Chest radiograph; Diagnostic Test: Lung ultrasound; Diagnostic Test: cell free DNA test
- Control group--Test population: Well Children Control Group-One for each child in groups A-C above, age matched for paired case.
  * Well children presenting for reasons other than respiratory diseases, and not symptomatic for TB.
  * Clinical and radiographic evaluation (if performed) NOT suggestive of TB, and NOT diagnosed or treated for TB during the follow-up period (minimum 8 weeks).
  * Divided into 2 subgroups based on presence or absence of LTBI (by Quantiferon Gold assay).
  Interventions: Diagnostic Test: Quantiferon Gold; Diagnostic Test: HIV serology; Diagnostic Test: cell free DNA test
- Presumptive pediatric TB cases-- Validation population: Inclusion criteria: Children ages 2 months to 14 years with symptomatic disease and suspicion of TB (based on Bolivian Ministry of Health guidelines).
  Exclusion criteria (prior treatment for TB in 12 mo, current treatment for TB, weight < 2.5 kg., instability, positive COVID-19 test) Study subgroups are determined in part based on the results of diagnostic tests and on clinical response.
  A. Confirmed TB
  * Symptomatic by case definition from the 2015 NIH Expert Panel
  * Positive culture or positive Xpert MTB/RIF from at least one sample.
  B. Unconfirmed TB-
  * Symptomatic and clinical/radiographic evaluation consistent with TB, by case definition from the 2015 NIH Expert Panel
  * Negative M. tuberculosis culture and negative Xpert MTB/RIF from all samples.
  C. Unlikely TB---
  * Symptomatic BUT clinical/radiographic eval does NOT meet criteria for Unconfirmed TB, per clinical definition-2015 Expert Panel
  * Negative culture and negative Xpert MTB/RIF from all specimens.
  Interventions: Diagnostic Test: Quantiferon Gold; Diagnostic Test: HIV serology; Diagnostic Test: Respiratory secretion culture (sputum or gastric aspirate_; Diagnostic Test: Chest radiograph; Diagnostic Test: Lung ultrasound; Diagnostic Test: cell free DNA test
- Control group--Validation population: Well Children Control Group-One for each child in groups A-C above, age matched for paired case.
  * Well children presenting for reasons other than respiratory diseases, and not symptomatic for TB.
  * Clinical and radiographic evaluation (if performed) NOT suggestive of TB, and NOT diagnosed or treated for TB during the follow-up period (minimum 8 weeks).
  * Divided into 2 subgroups based on presence or absence of LTBI (by Quantiferon Gold assay).
  Interventions: Diagnostic Test: Quantiferon Gold; Diagnostic Test: HIV serology; Diagnostic Test: cell free DNA test

INTERVENTIONS:
Diagnostic Test: Quantiferon Gold — Test for TB infection
Diagnostic Test: HIV serology — Test for HIV infection
Diagnostic Test: Respiratory secretion culture (sputum or gastric aspirate_ — TB culture by MODS
  Groups: Presumptive pediatric TB cases-- Test population; Presumptive pediatric TB cases-- Validation population
Diagnostic Test: Chest radiograph — Chest imaging test by traditional X ray
  Other Names: Chest X ray
  Groups: Presumptive pediatric TB cases-- Test population; Presumptive pediatric TB cases-- Validation population
Diagnostic Test: Lung ultrasound — Chest imaging test by ultrasound
  Groups: Presumptive pediatric TB cases-- Test population; Presumptive pediatric TB cases-- Validation population
Diagnostic Test: cell free DNA test — Blood test for TB infection

SUMMARY:
Pediatric tuberculosis (TB) continues to pose diagnostic challenges in low- and middle-income countries with high rates of TB disease, due to the well-described impact of paucibacillary disease in children, and current TB culture and polymerase-chain reaction tests are of limited usefulness due to cost, restricted availability, and poor sensitivity in specimens available from younger children. Our team of experts from Tulane, Johns Hopkins University, Universidad Peruana Cayetano Heredia, and Asociación Benéfica Prisma have confronted all of these challenges through more than 25 years of collaboration in Peru and Bolivia. Our goal is to directly address the challenges of TB in children by evaluating a new diagnostic approach developed by MPI Tony Hu at Tulane University using a CRISPR-mediated TB assay (CRISPR-TB) optimized to detect circulating Mycobacterium tuberculosis cell-free DNA (Mtb-cfDNA), and used to analyze cryopreserved serum in pilot studies from adults and children with presumptive TB, their asymptomatic household contacts, and a cohort of symptomatic children living with HIV (CLHIV) at high risk for TB. Results from symptomatic adult cohorts yielded a pooled sensitivity of 93%; specificity of 93%; positive predictive value of 95%; and negative predictive value of 92%. In limited pilot studies in CLHIV CRISPR-TBD results accurately identified all confirmed TB (13/13) and most children with unconfirmed TB (80%; 52/65). We propose to enroll 200 presumptive TB cases and an equal number of well control subjects in each of 2 study populations (test population and validation population) identified through clinics associated with the "Dr. Mario Ortiz Suarez" Children's Hospital in Santa Cruz, Bolivia. We will determine the distribution of cfDNA concentrations in peripheral blood in a "test population" composed of two age-based groups of children (2 months-6 years, 7-14 years) with respiratory disease grouped by likelihood of TB based on the NIH consensus case definitions (confirmed TB, unconfirmed TB, and unlikely TB) and in age-matched controls grouped by presence of latent TB infection (LTBI), with cfDNA measured serially in time among TB cases receiving antibiotic therapy. We will also validate standard ranges of quantitative cfDNA established for clinical subgroups of children with TB disease or LTBI in an independent validation cohort. An additional aim will determine the correlation between quantitative cfDNA and quantitative imaging-based TB scores based on evidence of disease in the lung, the primary target organ in TB disease, by (1) chest radiograph, measured by computer-aided analysis using the CAD4TB v7 system, and by (2) lung ultrasound, performed with a portable/low-cost probe assisted by machine learning algorithms for automatic interpretation. These biomarkers will be tested as potential cofactors that may be combined with cfDNA levels in peripheral blood, to improve the detection of TB disease in children. The results of this study will be the first step in a process to find a path to allow detection of the many "unconfirmed" TB cases and ideally make the diagnosis of pediatric TB in reach for low resource settings where it is so critically needed.

DETAILED DESCRIPTION:
Pediatric subject populations, enrollment, and follow-up: During the first two years of the study, a "test population" will be recruited for 18 months to establish quantitative cfDNA standards and ranges for each clinical outcome group, to assess predictive values for cfDNA levels as a biomarker of clinical outcome. We will characterize the dynamics of cfDNA levels in peripheral blood in two age-based groups of children (2 months-6 years ["younger children"], 7-14 years ["older children"]). A stratified analysis with these age-based subgroups is logical because the diagnostic test yield and clinical presentations are different in these groups.

For Aim 2 during years 3-4 of the study, a "validation population" will be recruited for 18 months to validate quantitative cfDNA standards and ranges for each clinical outcome group. Subject recruitment, informed consent, data collection, and study groups for analysis will be the same as for the "test population" in Specific Aim #1. Subjects in each study group will be stratified into age-based subgroups (2 months-6 years, 7-14 years). Serial levels of cfDNA will be assessed and characterized for children in the confirmed and unconfirmed TB groups, to validate normalization of cfDNA values with effective anti-TB therapy.

Table 1. Project Timeline

Initial enrollment and data/specimen collection will be done prior to initiation of TB treatment in the hospital or clinic setting. Inclusion criteria: Children ages 2 months to 14 years identified through the clinics and hospital wards of the "Dr. Mario Ortiz Suarez" Children's Hospital in Santa Cruz and presenting for evaluation for symptomatic respiratory disease and suspicion of tuberculosis will be eligible for enrollment (inclusion criteria based on Bolivian Ministry of Health guidelines for suspect cases of tuberculosis in children ). After screening for exclusion criteria (prior treatment for TB within the past year, current treatment for prevention of TB, weight < 2.5 kg., or clinical instability, positive COVID-19 diagnostic test) study staff will present the study verbally to the parents and provide a brochure with more detailed information designed for both parents and older. Parental informed consent and pediatric participant assent will be obtained. The study will include collection of specimens for diagnostic testing and clinical data as outlined below, but decisions on treatment for tuberculosis will be made by the attending physician who is not involved in the study. As the study groups for data analysis are determined in part based on the results of diagnostic tests performed and on clinical response to treatment, subjects will not be assigned to study groups on enrollment. Study group assignment (confirmed TB, unconfirmed TB, and unlikely TB) will be determined by the project biostatistician after the subject completes all study activities (see D.5. and D.7. study group assignment for criteria and sample size by group). As the Bolivian guidelines for pediatric TB allow for clinical evaluation of children with respiratory disease and only a few TB-related criteria, this recruitment strategy will enroll a population of suspect TB patients that will allow us to compare outcomes in "TB cases" (confirmed TB and unconfirmed TB) and in ill patients who do not meet NIH case definitions for unconfirmed TB (i.e., the unlikely TB group, see D7). This unlikely TB group will serve as "ill/respiratory disease controls", separate from the "well controls" group. On a weekly basis, well control subjects without respiratory symptoms and age-matched (+ 2 years) to suspected TB cases will also be recruited from community health clinics. Well controls will only have a single set of specimens, and no invasive specimens.

D.4. Bolivia study staff: Recruitment of study participants and specimen collection activities will be managed by a physician study coordinator, supervised by co-investigator Dr. Ramiro Cabrera, pediatric pulmonologist and regional consultant for pediatric tuberculosis in Santa Cruz. Clinical and patient related activities will be further overseen by PIs Richard Oberhelman (pediatric infectious diseases specialist) and Robert Gilman (ID specialist), as well as by ID specialists Jeffrey Tornheim and Lima-based Prisma site director Carlton Evans.

D.5. Primary Outcomes, Statistical Power, and Sample Size The primary outcome for Aim 1 is cfDNA levels for a) children with confirmed and unconfirmed TB ("TB cases"), b) children with unlikely TB (UTB), and c) well children (WC). Based on preliminary data, the mean cfDNA levels (and standard deviations) for these groups were 4.2 (4.0), 2.0 (3.2), and 1.1 (0.03), respectively. We hypothesize that TB children will have significantly higher serum concentrations of cfDNA than the UTB and WC groups. Statistical power and sample size: With a two-sided type I error is set at 0.05, statistical power set at 80%, 42 subjects per group are required to detect a significant difference between the TB and UTB children (based on the formulae by Hulley et al. ). Comparisons between the TB and WC group requires 13 children per comparison group. Based on data from current studies and local Ministry of Health (see D.7. below) we anticipate 135 TB cases per year (55 in 2 mo-6 yrs.; 80 in 7-14 yrs.), or approximately 200 TB cases per 18-month study period (for test population and validation population). We also anticipate 80 unlikely TB cases per year (40 in 2 mo-6 yrs.: 40 in 7-14 yrs.), or approximately 105 unlikely TB cases per 18-month study period (18 months each for test population and validation population recruitment). Subjects will be stratified into two age groups (2 months-6 years, 7-14 years). With 42 required TB cases per age group, our proposed sample exceeds the minimum requirements by 50% or more per age group. The enrollment targets here will provide flexibility in meeting recruitment goals and non-response rates.

D.6. Procedures and specimen collection. For hospitalized patients with suspected tuberculosis, enrollment, clinical evaluation, and sample collection are performed in the same room; for outpatients the process of clinical evaluation, gastric aspirate sampling will be performed in the consulting room of Pneumology clinic at the pediatric hospital and blood sampling will be collected in the clinical laboratory phlebotomy room. Follow-up specimen collection will be done through community clinics where patients receive their weekly allotment of TB medicines, with follow-ups at 1- and 2-weeks post treatment initiation. A 2-month follow-up visit in conjunction with a routine physician visit is scheduled, to allow for a later follow-up cfDNA biomarker specimen.

All participants under evaluation for TB will have procedures at the time of enrollment including:

* Medical history and clinical evaluation required to accurately assess each criterion that contributes to their subsequent assignment to TB outcome groups, based on the 2015 revised consensus criteria.
* Quantiferon-TB Gold In-Tube testing to detect immunologic evidence of tuberculosis (including latent infection [LTBI]) will be performed in our laboratory at Universidad Catolica, based on standard protocols
* HIV serology unless known to be HIV+, by Abbott Alere Determine HIV 1/2 (See D.8 Data analysis for analytical adjustments by HIV serostatus)
* COVID-19 PCR or antigen test-- suspect TB patients only. (If positive these subjects are excluded)
* Chest radiograph-- suspect TB patients only; not performed on well controls. AP and lateral views. Digital images processed in DICOM will be transmitted to Dr. Zimic's lab for analysis.
* Lung ultrasound-- suspect TB patients only; Not performed on well controls. Ultrasound examination is performed based on a standard protocol supervised by Dr. Fentress, imaging the chest in perpendicular planes in the midclavicular line anteriorly and posteriorly from apices to diaphragm, and in the midaxillary line from axilla to diaphragm, for a total of 12 views per participant. , ,
* Specimen collection for TB microbiology and PCR-- suspect TB patients only; not performed on well controls. All subjects with a work-up for suspected TB will have at least three sputum-equivalent specimens collected for TB microbiology and PCR analysis by Xpert MTB/RIF. Acceptable specimens include (1) gastric aspirates, (2) expectorated sputum (for older subjects who can produce sputum), or (3) string test specimens, conducted by our standard protocol. Specimens will be collected in the early morning prior to eating, and specimen collection times will be separated by at least 24 hours. In cases where parents or attending physicians only agree to two specimens, a third specimen will not be collected. Anti-TB treatment will be initiated when indicated by the physician following collection of the last specimen for TB microbiology.
* Microbiologic analysis for TB isolation and detection will be performed on specimens collected from suspect TB patients, including (1) Ziehl-Neelsen AFB smear, (2) TB culture, and (3) and TB PCR detection by Xpert MTB/RIF. TB cultures will use the MODS technique that we developed in Peru 8, 10
* Serum for cfDNA collected by venipuncture. We ship all serum cfDNA samples to Tulane by World Courier, on dry ice, and we aliquot all samples so half will be shipped and the other half stored at -80 C.

Participation by well control subjects will end after enrollment specimen collection and evaluations. TB treatment will be initiated for all subjects with presumptive TB disease, based on the attending physician's clinical opinion and based on Bolivian national TB treatment standards. Study participants with compatible disease and on anti-TB therapy will have the follow-up procedures listed at the times specified:

* Clinical evaluation (1 week, 2 weeks, and 2 months post enrollment and start of treatment)
* Serum for cfDNA and whole blood for CBC (1 week, 2 weeks, and 2 months post enrollment)
* For subjects on antituberculous therapy and not demonstrating improvement-repeat evaluation (per clinician decision at 2 weeks or 2 months post enrollment). Minimum 2 samples for smear, culture, and Xpert MTB/RIF (Gastric aspirates [by intubation/string test] or sputum)

TB culture techniques. Specimens collected will be cultured for M. tuberculosis using the Microscopic-Observation Drug-Susceptibility (MODS) Method.8 Standard volumes of each decontaminated specimen will be inoculated into modified Middlebrook 7H9 media and cultured in a sterile 24-well plate. Plates are placed in a plastic resealable bag, incubated at 37°C, and examined every other day for up to 30 days by inverted light microscopy. Presumptive TB isolates with cording are reported as positive and confirmed by IS 6110 PCR.

CRISPR-TBD assays: The circulating cfDNA will be extracted with Quick-cfDNA Serum & Plasma at the Hu lab at Tulane. CRISPR-TBDB requires an PCR-based target amplification prior to CRISPR-mediated fluorescent signal production, following procedures recently published by Huang et. al. 23 The CRISPR-TBDB data will be evaluated in silico analysis using SnapGene software (version 5.0.8) and by triplicate CRISPR-TBDB assays.

Chest radiograph and lung ultrasound studies and data processing. See Specific Aim #3 below.

D.7. Study group assignment. We will employ an observational study design with 5 study groups of children ages 2 months to 14 years, as detailed below. These are A) confirmed pulmonary TB, B) unconfirmed pulmonary TB, C) unlikely TB, D) well age-matched controls (which will be divided into 2 groups based on presence or absence of LTBI). Most children evaluated for TB and started on treatment as determined by the attending (non-study) physician will fall into groups A (approximately 10%) and B (60-65%), based on recent data. Groups A and B together are referred to here as "TB cases". Approximately 25-30% of subjects who meet entry criteria based on Bolivian guidelines but fail to meet the 2015 NIH guidance definition for confirmed or unconfirmed will be included as group C (unlikely TB), serving as an "other respiratory disease" comparison group. The estimated eligible population is based on data from the ongoing R21 study (for children aged 0-5 years) and on data from the Ministry of Health. Criteria for each study group and estimated number per group to be recruited per year during subject enrollment periods are:

A. Confirmed TB- estimated 65 subjects per year (15 in 2 mo. - 6 yr.; 50 in 7 - 14 yr.), defined as:

* Symptomatic at initial enrollment, defined based on the clinical case definition from the 2015 NIH Consensus Expert Panel 22 (Quantiferon Gold positive or negative).
* Positive M. tuberculosis culture or positive Xpert MTB/RIF from at least one biological sample.

B. Unconfirmed TB-estimated 80 subjects per year (40 in 2 mo. - 6 yr.; 30 in 7 - 14 yr.) defined as:

* Symptomatic at enrollment and clinical/radiographic evaluation consistent with TB, based on the clinical case definition from the 2015 NIH Consensus Expert Panel 22 (Quantiferon Gold positive or negative).
* Negative M. tuberculosis culture and negative Xpert MTB/RIF from all biological samples.

C. Unlikely TB--- 80 subjects per year (40 in 2 mo. - 6 yr.; 40 in 7 - 14 yr.), defined as:

* Symptomatic at enrollment BUT clinical/radiographic evaluation does NOT meet criteria for Unconfirmed TB, per clinical definition-2015 Expert Panel 22 (Quantiferon Gold positive or negative).
* Negative M. tuberculosis culture and negative Xpert MTB/RIF from all specimens. D. Well Children Control Group-One for each child in groups A-C above, age matched for paired case.
* Well children presenting for reasons other than respiratory diseases, and not symptomatic for TB.
* Clinical and radiographic evaluation (if performed) NOT suggestive of TB, and NOT diagnosed or treated for TB during the follow-up period (minimum 8 weeks).
* Divided into 2 subgroups based on presence or absence of LTBI (by Quantiferon Gold assay).

D.8. Data analysis. Subjects will be sorted at the time of data analysis based on diagnostic test results into "confirmed," "unconfirmed," and "unlikely" TB based on diagnostic test results and clinical evolution. Since most children under age 7 with TB disease do not have culture or Xpert confirmation, and unconfirmed TB cases are considered true cases for epidemiologic purposes, these groups will also be combined as "TB cases" for analysis. Subjects in each study group will be stratified into age-based subgroups (2 months-6 years, 7-12 years). For exploratory analyses, additional subgroups based on HIV serostatus will be conducted both including and excluding HIV+ subjects (HIV seroprevalence is extremely low in children in this population, so the impact of HIV status will likely be minimal). Sex will be considered as an independent variable in all analyses. Additionally, sex will be included as an interaction term against all primary predictor variables (time of observation, cfDNA level). Serial levels of cfDNA will be assessed and characterized for children in the confirmed and unconfirmed TB groups. Replicate cfDNA values will be standardized by modeling their average values against their corresponding concentrations using four-parameter logistic regression models. Mann Whitney U tests will be used for testing hypotheses comparing the TB case group with the three comparison groups (children with unlikely TB, well children with LTBI, and well children without LTBI). Exploratory analyses will compare outcomes (cfDNA level, TB risk scores) between the "gold standard" confirmed TB (culture or Xpert MTB-RIF positive) group and the unconfirmed (culture and Xpert negative) group. A Bonferroni correction factor will be applied to account for multiple testing over the age group strata.

For response to treatment analysis (Specific Aim 2), a positive response is defined as per 2015 clinical case definitions consensus paper, measured at 1 wk., 2 wks., and 2 mo. post enrollment, as either:

a) Response to antituberculosis therapy: clinical features suggestive of tuberculosis disease that were present at baseline have improved, and there is no new clinical feature suggestive of tuberculosis; OR (b) No response to antituberculosis therapy: clinical features suggestive of tuberculosis disease that were present at baseline have not improved or have worsened.

The analytical objective is to compare response differences in cfDNA levels over time. Generalized estimating equations (GEE) will be used to model response to treatment against time of observation and cfDNA level. An interaction term will be included in the GEE model to test whether temporal pattens in cfDNA levels differ by response type. Pairwise comparisons will be performed to compare cfDNA levels between the response groups at each time point. Weighted GEE models will be used to account for missing follow-up data. To assess time to positive treatment response, Kaplan Meier curves will be applied, including treatment response as a censoring variable and plotted against cfDNA levels (classified into tertiles) over time.

D.9 Specific Aim #3: Determine the correlation between cfDNA levels and quantitative TB disease risk score biomarkers determined by (1) chest radiograph, measured by computer-aided analysis, and by (2) lung ultrasound, performed with a portable/low-cost probe and assisted by machine learning algorithms for automatic interpretation without requiring a radiologist. These biomarkers will be tested as potential cofactors that may combine with cfDNA levels in peripheral blood, to improve the detection of TB disease in children. As a secondary goal, we will examine chest radiograph and lung ultrasound findings using artificial intelligence algorithms for interpretation, to explore potential associations between cfDNA and imaging biomarkers. The fact that imaging findings are the most concrete evidence of disease available among the many "soft" diagnostic criteria validates this exploratory analysis in spite of limited sensitivity and specificity. If presence of lung pathology by imaging among children with TB correlates with cfDNA level, this would be a finding with immense clinical utility for health professionals in LMICs. However, interpretation of chest radiographs is arguably the most challenging component of TB diagnostic criteria since it requires sophisticated, expensive equipment and expert staff, both technicians for data collection and health professionals for interpretation. We propose a multifaceted approach to the analysis of imaging data, utilizing two unconventional approaches that are supported in the medical literature, i.e. 1) lung ultrasound as a radiation-free alternative to chest radiograph that is generally more portable, with several low-cost, portable platforms; and 2) utilization of automated interpretation of both chest radiographs and LUS, using machine learning computer-aided design (CAD) technology. Of several CAD technologies marketed for interpretation of chest radiographs in patients with tuberculosis ages 15 and higher, only one is extensively validated and CE certified in the European Union for use in children ages 4 and up-the Delft Imaging CAD4TB platform. , , CAD4TB processes DICOM images by chest radiograph to produce a score from 0 to 100 to assess probability of active TB, as well as a heat map image to indicate sections of the lung with TB-related pathology (see Fig. 7). The CAD4TB software and technical support for this study will be donated by Delft Imaging (see letter of support). In addition, Dr. Mirko Zimic will use machine learning approaches used to develop algorithms for pediatric pneumonia by LUS to develop a similar strategy for pediatric TB. Both the CAD4TB platform and the Zimic LUS algorithm will produce a TB risk score that can be compared to radiologist's interpretations, and both the AI-based risk scores and traditional risk scores will be correlated with cfDNA levels.

All ultrasound scans will be performed by trained staff using a General Electric VIVID i BT12 with a high frequency linear probe. The sonographer will record the presence and location of abnormal ultrasound findings as per Fentress et. al. 16 We will record at least one video from each sonographic view to allow for external review after scanning, for at least 12 ultrasound videos per participant.

D. 10. Imaging interpretation and analysis: Chest radiograph outcomes will be recorded in two formats:

1. Radiographs will be reviewed independently by two pediatric radiologists who will note the presence or absence of specific findings suggestive of PTB, as defined by the 2015 expert panel. 22 These findings include lymphadenopathy, air space opacification, nodules, and pleural effusions. Reports from the radiologists will be compared to determine congruency with "consistent with tuberculosis" as per 2015 clinical criteria. In cases where the determination is discordant, a third radiologist will make a determination. Radiologists will record findings and severity based on a standard scale, to produce a risk score for analysis.
2. DICOM images will be evaluated using the CAD4TB v7 program, using published procedures, to generate a TB risk score and heat map image of the lungs.

Conventional chest X ray scores are determined by the number of findings checked as positive (out of a total n =8 possible findings) based on the NIH consensus paper CXR template. CAD4TB is trained on independent annotated datasets to recognize features of TB, and it outputs a score 0-100 which indicates the probability of TB. An abnormality heatmap is also generated to indicate regions of the lung detected as abnormal. The analysis plan includes three factors: Conventional X-ray or CAD4TB score (ordinal response variable), time of observation, and cfDNA level. The analytical objective is to test for significant differences between CAD4TB score values and cfDNA levels over time. GEE will be used to model CAD4TB scores against time and cfDNA level. An interaction term will be used to test whether temporal trends in cfDNA levels differ by CAD4TB score. Pairwise comparisons will be used to test for significant differences between cfDNA levels and CAD4TB scores at each time point. Weighted GEE models will be used to account for missing follow-up data. 31

Lung ultrasound (LUS) outcomes will similarly be evaluated by both conventional and automated machine learning approaches. All saved ultrasound images will be reviewed by a lung ultrasound expert blinded to the participant's clinical data. When there is disagreement between the field sonographer's interpretation and the blinded LUS expert, this will be adjudicated by a second blinded ultrasound expert. LUS images will be visually assessed and classified as positive or negative for TB based on 2015 expert panel-defined lung findings for chest radiographs applied to LUS. An artificial convolutional neural network (CNN) based on lung ultrasound images will be trained for prediction of TB by methods previously published by Zimic et. al.,22, 23 according to the gold standard classification based on NIH criteria and chest radiographs. In previous studies, we developed a CNN for TB recognition in MODS cultures which achieved 96% accuracy, 96% sensitivity and 96% specificity, demonstrating that CNNs could assist or replace personnel for the automated diagnosis of TB.22, 23 The training of the proposed CNN will be done using the Caffe and Tensorflow frameworks because their speed and modularity. The system will be developed in Python using OpenCV libraries in the detection step. Every frame of each LUS video will be labelled manually by the expert, to determine if it has evidence of TB lesions. We will use a LeNet CNN variant model, relying on two convolutional layers, each one followed of pooling operations like sub-sampling that will account for translation invariance. The combination of the aforementioned layers is expected to give a total of 60K learnable parameters. With approximately 280 children expected to be enrolled in the first two years, each with 1-minute videos extracted from LUS at 30 frames per second (1,800 frames), we will have a total of 504,000 images. Using standard data augmentation, we expect to at least have 4x106 images for an adequate CNN training. Multiple logistic regression analyses will be used to model the gold-standard TB classification TB, including as predictors the cfDNA level and ultrasound CNN score, adjusting for age and sex.

LUS analysis will be performed with methodologies similar to those used for CXR, adapted for LUS-based outcomes. LUS score will be adapted from the NIH consensus paper for CXR and will consist of a combination of the quantitative number of findings checked as positive (out of a total n=5: consolidation, small subpleural consolidation, cavity, pleural effusion, and miliary pattern) and the number and location of abnormal lung regions, incorporated into a logistic regression model. LUS will also be interpreted as "consistent with TB" or "not consistent with TB", based on the same criteria used for CXR in the NIH consensus paper. The GEE-based approach described above for CXR will also be applied to analysis of LUS data.

ELIGIBILITY:
Inclusion Criteria:

* Children presenting for evaluation for symptomatic respiratory disease and suspicion of tuberculosis will be eligible for enrollment (inclusion criteria based on Bolivian Ministry of Health guidelines for suspect cases of tuberculosis in children

Exclusion Criteria:

* prior treatment for TB within the past year,
* current treatment for prevention of TB,
* weight < 2.5 kg., or
* clinical instability,
* positive COVID-19 diagnostic test

Ages: 2 Months to 14 Years | Sex: All
Age Groups: Child
Study Population: Children from clinic population in Santa Cruz Bolivia
Sampling Method: Non-Probability Sample
Enrollment: 1220 (Estimated)
Dates: Start 2024-04-15 (Actual); Primary Completion 2027-10 (Estimated); Study Completion 2028-10 (Estimated)

PRIMARY OUTCOMES:
Cell free DNA level | Baseline and 2 months post treatment for TB cases on therapy
  Cell free DNA level

SECONDARY OUTCOMES:
CAD4TB score | At presentation for case grou
  Artificial intelligence interpretation of chest radiograph for likelihood of TB

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital de Ninos "Mario Ortiz Suarez", Santa Cruz, Bolivia

IPD SHARING:
Plan to Share IPD: Undecided